CLINICAL TRIAL: NCT06572293
Title: Nurse-Led Individualized Follow-Up Intervention Versus Regular Physician-Led Visits in Nasopharyngeal Carcinoma: A Phase III Randomized, Controlled Trial
Brief Title: Effect of Nurse-Led Individualized Follow-Up Intervention on Patients With Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiaojuan Guo, M.D, Professor, Fujian Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-6-6
Record Dates: First submitted 2024-07-31; First posted 2024-08-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Nurse-Led Individualized Follow-Up; post-radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Nurse-led follow-up
  Interventions: Behavioral: Nurse-led intervention
- Control (No Intervention): Physician-led follow-up

INTERVENTIONS:
Behavioral: Nurse-led intervention — Nurse-led intervention involves patient education, collecting Patient Reported Outcomes (PRO) and evaluating them by specialists nurses, as well as navigating patients to services that can assist with their symptoms. During three-five planned appointments, the nurse will talk with you about adjusting to life after complete the radiotherapy of nasopharyngeal carcinoma, including symptoms of relapse and how to deal with them.In the first year, PROs will be collected every six months on recurrences and late effects, and thereafter every 12 months. PRO will be administered to patients for three years after the nurse appointments are finalized.
  Arms: Intervention

SUMMARY:
The incidence of nasopharyngeal carcinomas (NPCs) is highly unbalanced around the globe, primarily concentrated in East and Southeast Asia.There is no well-conducted, larger randomized controlled trials (RCT) outlining a gold standard for follow-up programs ensuring early detection of recurrence, good management of symptoms and cost-effectiveness. The primary aim of this randomised, controlled trial is to test whether a nurse-led individually tailored symptom management program will significantly reduce reported symptoms among NPC patients following primary treatment compared to physician-led scheduled follow-up. Additionally, the investigators will assess patient activation (self-management), anxiety, depression, fear of recurrence, work abilities, recurrence times, changes in health behavior, and health care utilization and costs for the two arms of the study.

A nurse-led education program focused on symptom management is provided to patients, along with an electronic platform to report symptoms to nurses and support in symptom management.

DETAILED DESCRIPTION:
It is planned to recruit 250 primary NPC patients from Fujian Cancer Hospital's Oncology Departments during an 18-month period, after completing the chemoradiotherapy for NPC. You will participate in a five-year study in which you are randomly assigned to either the nurse-led intervention or the physician-led intervention. Regardless of group assignment, you will follow the national nasopharyngeal carcinoma screening program.

Both the control and intervention arms will use questionnaires, clinical databases, and national registers to collect data for 5 years after inclusion both in the control and intervention groups. The primary and secondary outcomes are measured using questionnaires in both groups, whereas Patient Reported Outcomes (PRO) are collected only in the intervention group. Relapsed patients will not be asked to complete the remaining outcome questionnaires or PROs since they quit the follow-up program to pursue recurrent treatment. If PROs reveal a need, or if the patient requires consultation, the nurse or project physician will be consulted.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent;
2. Have completed radiotherapy treatment for loco-regional nasopharyngeal carcinoma without clinical sign of distance metastatis;
3. Aged 18 years and above;
4. Expected survival ≥6 months;
5. Read, understand Chinese characters and speak Mandarin.

Exclusion Criteria:

1. Previous history of other malignancies, mental illness or cognitive impairment (MMSE score < 27 points);
2. Unstable medical or psychiatric conditions
3. Inability to communicate effectively in mandarin
4. Pregnant women or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life score (EORTC QLQ C30) | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Quality of life score was calculated according to the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ C30), the range is 0-100, higher scores mean a worse outcome.
Quality of life score QLQ-HN35 | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Quality of life score was calculated according to the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire QLQ-HN35, the range is 0-100, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes in knowledge, skill, and confidence for self-management | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Patient Activation Measure (PAM), interval-level scale from 0-100 that correlates to one of four levels of patient activation. PAM Levels 1 and 2 indicate lower patient activation, while PAM Levels 3 and 4 indicate higher patient activation.
Changes in anxiety | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Generalized Anxiety Disorder (GAD-7),the range is 7-28, higher scores mean a worse outcome.
Changes in self-management | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  The Health Education Impact Questionnaire (heiQ), the range is 40-160, higher scores mean a better outcome.
Changes in fear of recurrence | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Concerns About Recurrence Questionnaire (CARQ-4),the range is 0-40, and a higher score represents higher fear of recurrence.
Changes in Depression | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  The Patient Health Questionnaire (PHQ-9),the range is 0-27, higher scores mean a worse outcome.
Changes in work ability | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Work Ability Index (WAI), range 7-49, a higher score indicated better work ability

CONTACTS AND LOCATIONS:
Overall Officials: Qiaojuan Guo, Dr., Principal Investigator — Fujian Cancer Hospital